CLINICAL TRIAL: NCT06091293
Title: Narrative Intervention for Long COVID-19 (NICO) Research Study
Brief Title: Narrative Intervention for Long COVID-19 (NICO)
Acronym: NICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0701
Record Dates: First submitted 2023-10-18; First posted 2023-10-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Long COVID; Long Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: This study has one arm. All participants will receive the NICO intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NICO (Experimental): The NICO intervention includes components of narrative-informed interventions, brief solution-focused therapy, and medical social work case management to examine adjustment to illness for people living with Long COVID.
  Interventions: Behavioral: Narrative Intervention for Long COVID-19 (NICO)

INTERVENTIONS:
Behavioral: Narrative Intervention for Long COVID-19 (NICO) — The NICO intervention was delivered by a licensed psychotherapist asynchronously over a 3 month time period.

SUMMARY:
This T1 proof of concept trial is designed to test the Narrative Intervention for Long COVID-19 intervention.

DETAILED DESCRIPTION:
People living with COVID19 Long Haul Syndrome frequently experience high symptom burden and problems performing basic activities of daily living. COVID19 has impacted mental health not only for people directly affected by the pandemic, including people who are living with COVID19 Long Haul Syndrome, but also those affected indirectly, putting further strain on the mental health system, which was already under stress.

Understanding the experience of COVID 19 Long Haul Syndrome that can inform innovative and impactful ways to improve living with COVID19. Mental health providers are in high demand with an increase in burnout. One study reported 1/3 of mental health providers have experienced severe burnout since the onset of the pandemic. There are nursing staff shortages across the US, especially in rural areas. Shortages also occur within social work staff globally. There is a need to design innovative, interdisciplinary, and less time-intensive interventions to help those living with chronic illness. More people living longer with different types of illnesses and staffing shortages make traditional talk therapy interventions more challenging to deliver to more people.

This study has two specific aims:

Aim 1: Establish the acceptability and feasibility of an asynchronous narrative intervention for people living with long haul COVID19.

Aim 2: Explore themes of illness narratives of people living with long haul COVID19

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Long COVID
* Have access to email weekly
* Between the ages of 18-89 years old

Exclusion Criteria:

* Conflicting research study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Personal Health Questionnarrie- 8 item (PHQ8) | Baseline and 3 months
  Measurement of depression widely used in clinical and research settings

SECONDARY OUTCOMES:
Generalized Anxiety Disorder- 7 item (GAD7) | Baseline and 3 months
  Measurement of anxiety widely used in clinical and research settings

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Johnson, PhD, LCSW, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No